CLINICAL TRIAL: NCT05219422
Title: Improving the Implementation of Evidence-based Drug Prevention Programs in Schools
Brief Title: Testing ALERT With GTO in Middle Schools
Acronym: GTO-ALERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Matthew Chinman, Senior Behavioral/Social Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-0121-AM01
Record Dates: First submitted 2021-09-14; First posted 2022-02-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants from 42 schools will be randomized to received Project ALERT, Project ALERT + Getting to Outcomes, or waitlist control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Project ALERT only (Active Comparator): Some schools will be randomized to receive Project ALERT only for 3 years starting fall 2022.
  Interventions: Behavioral: Project ALERT
- Project ALERT plus GTO (Active Comparator): Some schools will be randomized to receive Project ALERT plus Getting to Outcomes for 3 years starting fall 2022.
  Interventions: Behavioral: Project ALERT; Behavioral: Getting to Outcomes
- Status quo (No Intervention): Some schools not receive either Project ALERT or Project ALERT plus GTO until year 3 of the study.

INTERVENTIONS:
Behavioral: Project ALERT — 14 session drug prevention program for 7th and 8th grade youth.
  Arms: Project ALERT only; Project ALERT plus GTO
Behavioral: Getting to Outcomes — The Getting To Outcomes (GTO) implementation support intervention provides technical assistance, training, guides, and tools to improve community-based practitioners capacity to complete tasks associated with implementing an EBP, which in turn leads to improved implementation fidelity.
  Arms: Project ALERT plus GTO

SUMMARY:
To test the efficacy of Project ALERT with the support enhancement tool, Getting To Outcomes.

DETAILED DESCRIPTION:
This study combines two programs that have been developed by RAND researchers: Project ALERT (PA) and Getting to Outcomes (GTO). Project ALERT is a widely used drug prevention program for middle school youth. Though it has an evidence-base for effectiveness, the program (like most evidence-based programs in schools) is not run with adequate fidelity representing a large gap between what is developed and tested for effectiveness and what is used in actual practice. Thus, the study will conduct an updated randomized controlled trial of PA and test GTO as a tool to increase adoption and adequate fidelity of the program in schools. GTO's previous evidence suggests it could be effective in public schools, yet this remains an empirical question. A successful demonstration of PA and GTO could fundamentally transform evidence-based prevention's delivery, reach, and thus impact, in the US.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for student participants: all students in 7th grade, primarily aged 12-14, attending school at one of the enrolled schools in the study.
* Eligibility for school staff participants: all educators interested in enrolling in the study at each of the enrolled schools.

Exclusion Criteria:

* Not meeting eligibility criteria

Note: the age range is from 11 to 70 to account for both the student AND teacher populations.

Ages: 11 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Student alcohol and drug behavior | Changes assessed for past year use at each follow-up point from baseline
  Alcohol and drug use will be assessed for alcohol, cigarettes, marijuana, e-cigarettes, prescription opioids, and heroin (lifetime, past month, past year use), allowing us to evaluate program effects on ever, past month, and weekly use. We will assess marijuana and nicotine using items to capture nuanced products (e.g., JUUL/vape pens) and include combinations of marijuana/nicotine products to assess co-use, such as using a vaporizer to vape both nicotine e-liquid and cannabis oil. For alcohol, we will ask questions that allow us to construct 3 alcohol misuse scales: (1) alcohol-related consequences (sum of 5 dichotomous questions on: getting sick, getting in a physical fight, getting in trouble at school, getting in trouble at home, doing something he/she later regretted); (2) high-risk drinking (sum of 3 dichotomous variables: binge drinking in the past month, polydrug use of alcohol and marijuana in the past year, weekly drinking); and (3) overall misuse (sum of above 8 variables).
Student pro-substance use risk factors on consequences | Changes assessed for past year consequences of use at each follow-up point from baseline
  Beliefs about the short- and long-term consequences (positive and negative). Measures come from the Project ALERT survey posted on the Project ALERT website and utilized in the 4 prior RCTs of Project ALERT.
Student resistance self-efficacy | Changes assessed for past year self-efficacy use at each follow-up point from baseline
  Resistance self-efficacy from the Project ALERT survey measures avoiding use of all 6 drugs in risky situations. Measure is posted on the Project ALERT website and utilized in the 4 prior RCTs of Project ALERT.
Student pro-substance use risk factors on perceived norms | Changes assessed for past year perceived peer use at each follow-up point from baseline
  Normative beliefs about the prevalence of use and its acceptability to others, including peers and parents. Measures come from the Project ALERT survey posted on the Project ALERT website and utilized in the 4 prior RCTs of Project ALERT.
Student pro-substance use risk factors on expectancies | Changes assessed for past year use at each follow-up point from baseline
  Expectations of drug use in the next 6 months. Measures come from the Project ALERT survey posted on the Project ALERT website and utilized in the 4 prior RCTs of Project ALERT.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Chinman, PhD, Principal Investigator — RAND; Eric Pedersen, PhD, Principal Investigator — University of Southern California
Locations (1):
- Los Angeles Unified School District, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website that contains outcomes measures — https://www.projectalert.com/

DOCUMENTS (1):
  • Informed Consent Form (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT05219422/ICF_000.pdf